CLINICAL TRIAL: NCT03289273
Title: REFINE: Regorafenib Observational Study in Hepatocellular Carcinoma
Brief Title: Observational Study to Evaluate, Under Real-world Practice Conditions, the Safety and Effectiveness of Regorafenib in Patients Diagnosed With Unresectable Hepatocellular Carcinoma (uHCC)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19244; EUPAS20981 (Registry Identifier: EMA)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Liver Neoplasms
Keywords: Liver cancer; unresectable hepatocellular carcinoma; real-world practice conditions; safety and effectiveness; management and treatment of liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- uHCC patients treated with regorafenib: Patients with a confirmed diagnosis of uHCC and for whom a decision to treat with regorafenib has been made (by the treating physician)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — As per the treating physicians discretion

SUMMARY:
Observational study to evaluate, under real-world practice conditions, the safety and effectiveness of regorafenib in patients diagnosed with unresectable hepatocellular carcinoma (uHCC)

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of unresectable HCC
* Physician-initiated decision to treat with regorafenib (prior to study enrollment)

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Past treatment with regorafenib

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Source population of the study are patients with unresectable hepatocellular carcinoma. Patients with this condition are mostly managed at specialist centers and cancer hospitals. The participation of these specialized centers in the study is going to ensure the representativeness of the study population. Physicians will be asked to sample consecutive patients whenever possible to avoid selection bias and thus increase the likelihood of representativeness.
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment emergent adverse events (TEAEs) leading to dose modifications (including reductions, interruptions and permanent discontinuation) | Up to 24 months
  The primary endpoint is the safety of regorafenib in patients with uHCC, defined as the frequency of documented TEAEs, including serious adverse events (SAEs).
  Safety will be assessed in all patients who receive at least one dose of regorafenib regardless of prior treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  Overall survival (OS) is defined as the time (days) from the start of regorafenib treatment to the date of death, due to any reason. Patients alive or lost to follow-up at the time of analysis will be censored at their last date of follow-up
Progression-free survival (PFS) | Up to 24 months
  Progression-free survival (PFS) is defined as the time (days) from the start of regorafenib treatment to the date of first observed disease progression (radiological or clinical, whichever is earlier) or death due to any cause, if death occurs before progression is documented
Time to progression (TTP) | Up to 24 months
  Time to progression (TTP) is defined as the time (days) from the start of regorafenib treatment to the first documented disease progression
Best overall tumor response (ORR) | Up to 24 months
  Best overall tumor response (ORR) will be defined according to investigator-assessed data according to local standard
Duration of regorafenib treatment | Up to 24 months
  Duration of regorafenib treatment, defined by the time interval from the start of regorafenib treatment to the day of permanent discontinuation of regorafenib (including death)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (17):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - St. Joseph´s Hospital and Medical Center, Phoenix, Arizona
  - University of Florida Health, Gainesville, Florida
  - University of Louisville - Clinical Trials Unit, Louisville, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers University, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - C.R.Wood Cancer Center, Glen Falls Hospital, Glens Falls, New York
  - University of Cincinatti, Cincinnati, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Many locations, Multiple Locations, Argentina
- Many locations, Multiple Locations, Austria
- Many locations, Multiple Locations, Belgium
- Many locations, Multiple Locations, Canada
- Many locations, Multiple Locations, China
- Many locations, Multiple Locations, Denmark
- Many locations, Multiple Locations, Egypt
- Many locations, Multiple Locations, France
- Many locations, Multiple Locations, Greece
- Many locations, Multiple Locations, Italy
- Many locations, Multiple Locations, Japan
- Many locations, Multiple Locations, Netherlands
- Many locations, Multiple Locations, Russia
- Many locations, Multiple Locations, Saudi Arabia
- Many locations, Multiple Locations, South Korea
- Many locations, Multiple Locations, Spain
- Many locations, Multiple Locations, Sweden
- Many locations, Multiple Locations, Taiwan
- Many locations, Multiple Locations, Thailand
- Many locations, Multiple Locations, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/